CLINICAL TRIAL: NCT04956107
Title: Psychological Distress in Colorectal Cancer Patients Following Surgery With Either HIPEC or Pelvic Exenteration
Brief Title: Psychological distREsS hipEc oR pelVic Exenteration
Acronym: PRESERVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Karolinska University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Preserve
Record Dates: First submitted 2021-06-28; First posted 2021-07-09 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-11

CONDITIONS: Colo-rectal Cancer
Keywords: cytoreductive surgery; hyperthermic intraperitoneal chemotherapy; pelvic exenteration; adverse effects; psychological distress; anxiety; depression; fear of cancer recurrence; cognitive dysfunction; quality of life
MeSH Terms: conditions — Colonic Neoplasms; Anxiety Disorders; Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIPEC cohort: Patients undergoing cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) for colorectal cancer with peritoneal metastases
- PE cohort: Patients undergoing pelvic exenteration (PE) for colorectal cancer with involvement of the urinary bladder

SUMMARY:
The purpose of this study is to describe type and extent of psychological distress (adverse effects) in patients undergoing surgery for colorectal cancer with peritoneal metastases and after surgery for colorectal cancer with involvement of the urinary bladder.

DETAILED DESCRIPTION:
After being informed about the study all patients giving written informed consent will be distributed a questionnaire asking questions on depression, anxiety, self-reported cognitive issues, sleep issues, quality of life and 'fear of cancer recurrence'. All these aspects will be investigated using validated questionnaires.

Once the investigators have the preliminary results (type and extent of psychological distress developed after CRS+HIPEC or PE) the investigators plan to conduct a workshop. In this workshop experts in different areas regarding psychological distress, project leaders, professor from the 'National Center of Late Adverse Effects after Cancer in Pelvic Organs' (Denmark) and patients will participate. With the input of experts and patients, a treatment strategy will be developed, and also an assessment will be made concerning which patients are likely to benefit from treatment by these experts, and which patients could potentially benefit from counselling by their general practitioner or via self-helping tools at home. The investigators plan to conduct this workshop autumn 2021 and start counselling spring 2022.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone intended curative CRS+HIPEC for peritoneal metastases originated from colorectal cancer (HIPEC cohort) according to national Danish guidelines
* Patients who have undergone intended curative total or anterior pelvic exenteration (PE cohort) for advanced or recurrent colorectal cancer according to national Danish guidelines

Exclusion Criteria:

* Patients under 18 years
* Patients not speaking Danish or Swedish, respectively, in Denmark and Sweden
* Patients unable to give informed consent
* Patients undergoing CRS+HIPEC or PE for cancers others than CRC
* Terminally ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will prospectively include patients who have undergone surgery at Aarhus University Hospital, Karolinska University Hospital, Stockholm, and Skåne University Hospital, Malmö. Inclusion in Denmark will start February 2021 and in Sweden Summer 2021. Inclusion period is 15 months.
  The HIPEC cohort will be established as a cross-sectional study. For newly operated patients, inclusion will happen shortly after surgery with prospective questionnaire follow-ups at 3, 6 and 12 months after inclusion. For patients who have undergone CRS+HIPEC more than 3 months ago, initial inclusion can take place at 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Patients in the PE cohort will be included shortly after surgery with follow-up at 3 months, 6 months and 12 months after surgery.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Development of depression after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery
  Descriptive analysis will be done using the following questionnaire: PHQ-9 (patient health questionnaire)
Development of anxiety after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery
  Descriptive analysis will be done using the following questionnaire: GAD-7 (general anxiety disorder)
Development of cognitive dysfunction after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery
  Descriptive analysis will be done using following the questionnaire: Items regarding cognitive functioning from the EORTC item library
Development of sleeping issues after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery
  Descriptive analysis will be done using following the questionnaire: ISI (insomnia sleep index)
Development of fatigue after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery
  Descriptive analysis will be done using following the questionnaire: FACIT V4 (fatigue scale)
Development of ´fear of cancer recurrence' after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery
  Descriptive analysis will be done using following the questionnaire: Fear of cancer recurrence - SF

SECONDARY OUTCOMES:
Risk factors associated with developing psychological distress | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Univariate and multivariate regression analysis will be performed to identify potential risk

CONTACTS AND LOCATIONS:
Overall Officials: Rogini Balachandran, MD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Department of Surgery, Aarhus University Hospital, Aarhus, Denmark
- Sweden (2):
  - Department of Surgery, Karolinska University Hospital, Solna, Stockholm County
  - Department of Surgery, Skånes University Hospital, Malmö, Malmo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balachandran R, Thaysen HV, Christensen P, Zachariae R, Iversen LH. Biopsychosocial Late Effects After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy for Peritoneal Metastases from Colorectal and Appendiceal Cancer: A National Prospective Cohort Study. Ann Surg Oncol. 2024 Mar;31(3):1959-1969. doi: 10.1245/s10434-023-14618-6. Epub 2023 Dec 21. PMID 38127212